CLINICAL TRIAL: NCT06834516
Title: Early Feasibility Data Collection Using ClearSight on Children Less Than Two Years Old
Brief Title: ClearSight Baby Cuff
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-11
Record Dates: First submitted 2025-01-23; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- All study subjects: All study subjects will receive the ClearSight noninvasive finger cuff on one finger.
  Interventions: Device: ClearSight baby cuff

INTERVENTIONS:
Device: ClearSight baby cuff — Noninvasive device for continuous blood pressure monitoring

SUMMARY:
A prospective, single arm data collection study evaluating a prototype ClearSight finger cuff in pediatric patients.

DETAILED DESCRIPTION:
A prospective, single arm data collection study evaluating a prototype ClearSight finger cuff in pediatric patients under 2 years old

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age < 2 years
3. Availability of a standard blood pressure measurement as part of standard of care

Exclusion Criteria:

1. Any significant disfigurement or prior injury to a participant's finger that is intended to be used for monitoring with the prototype finger cuff
2. Inability to place finger cuffs appropriately due to subject anatomy, condition, or obstructive paraphernalia
3. Known sensitivities to system materials
4. Broken or open skin located at the site of the finger cuff
5. Proven left-right difference in blood pressure
6. Cardiac problems that can cause a difference in blood pressure between the two arms, including aortic coarctation
7. Extreme contraction of the smooth muscles in the arteries and arterioles of the lower arm and hand, such as may be present in patients with Raynaud's disease

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects will be less than 2 years of age with blood pressure monitoring as part of routine care.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Proper cuff fit | 30 minutes of monitoring with study devices during scheduled surgery procedure
  The cuff fits properly on the participant's finger in at least 90% of total number of participants. Proper Fit is defined as complete overlap of the hook and loop areas attached to the cuff and the securement flap.
Cuff remains properly fitted for the duration of the study measurement | 30 minutes of monitoring with study devices during scheduled surgery procedure
  The cuff remains properly fitted for the duration of the study measurement for at least 90% of total number of participants.
Measurement with monitor started without errors | 30 minutes of monitoring with study devices during scheduled surgery procedure
  A measurement can be started without the monitor producing errors and a blood pressure waveform is measured in at least 60% of the attempts, unless the monitor is warning for vaso-constriction.
Measurement stability within 10 mins | 30 minutes of monitoring with study devices during scheduled surgery procedure
  The automatic physiological calibration (Physiocal) stabilizes to intervals ≥ 30 beats within 10 minutes in at least 60% of the attempts, indicating measurement stability unless the monitor is warning for vaso-constriction.
Early feasibility accuracy | 30 minutes of monitoring with study devices during scheduled surgery procedure
  For systolic blood pressure and diastolic blood pressure the mean value of the errors of all individual paired determinations of the ClearSight versus reference blood pressure shall be within or equal to ±5 mmHg, with a standard deviation, no greater than 8 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Abdelnour, MS, BSN, Study Director — Edwards Lifesciences
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, Netherlands, Netherlands

IPD SHARING:
Plan to Share IPD: No